CLINICAL TRIAL: NCT05934162
Title: Efficacy and Mediators of Change of Cognitive-behavior Therapy for PTSD: a Randomized Controlled Trial
Brief Title: Efficacy of Internet-delivered Cognitive-behavior Therapy for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Bragesjo, Clinical psychologist, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-02866-01
Record Dates: First submitted 2023-06-26; First posted 2023-07-06 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; therapist-guided treatment; internet delivered treatment; digital treatment; therapist-assisted treatment; prolonged exposure; trauma focused CBT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded assessors are used Participants know that are given a CBT treatment for PTSD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist-supported internet delivered prolonged exposure (Experimental): Therapist-supported internet delivered prolonged exposure comprising psychoeducation about PTSD, controlled breathing, imaginal exposure including processing, in vivo exposure and relapse prevention. The treatment will be delivered in a digital platform for ten weeks. Participants will have access to a therapist that will guide them through treatment in a text based format.
  Interventions: Behavioral: Therapist-supported internet-delivered prolonged exposure
- Therapist-supported CBT (Active Comparator): Therapist-supported CBT internet-delivered treatment comprising psychoeducation about PTSD, relaxation techniques and relapse prevention. . The treatment will be delivered in a digital platform for ten weeks. Participants will have access to a therapist that will guide them through treatment in a text based format.
  Interventions: Behavioral: Therapist-supported internet-delivered CBT

INTERVENTIONS:
Behavioral: Therapist-supported internet-delivered prolonged exposure — 10 weeks of therapist-supported internet-delivered prolonged exposure
  Arms: Therapist-supported internet delivered prolonged exposure
Behavioral: Therapist-supported internet-delivered CBT — 10 weeks of therapist-supported internet-delivered CBT
  Arms: Therapist-supported CBT

SUMMARY:
The goal of this clinical trial is to compare therapist-guided internet delivered prolonged exposure to an active control condition( therapist-guided internet delivered cognitive behavioral therapy containing relaxation techniques) for post-traumatic stress disorder.

The objective with this study is to investigate efficacy, mechanisms of change and cost effectiveness of therapist-guided internet delivered prolonged exposure.

Adult patients with post-traumatic stress disorder will be randomly assigned to receive either 10 weeks of therapist-guided internet delivered prolonged exposure or therapist-guided internet delivered cognitive-behavioral therapy containing relaxation.

DETAILED DESCRIPTION:
PTSD is a debilitating psychiatric disorder strongly linked to subsequent psychiatric and medical problems. Trauma-focused cognitive behavioral therapy (CBT-T) such as prolonged exposure is an effective treatment for PTSD and is recommended in most clinical guidelines as first-line treatment but is seldom available in regular care. A possible solution to significantly improve access to evidence-based treatment would be the use of remotely delivered digital intervention. Preliminary research shows that therapist-guided internet delivered to be effective and safe, but studies have typically excluded patients with severe PTSD.

Before this type of treatment can be offered in regular care in Sweden, it needs to be further evaluated also with psychiatric patients suffering from severe PTSD. If therapist-guided internet delivered prolonged exposure would be found to effective, this project has the potential to be the first step towards implementation of a novel, superior and more cost-effective mode of treatment delivery for adults with PTSD in regular Swedish health care.

The study is a single-blind, parallel-group superiority randomized controlled trial with 284 patients (142 per arm) that will compare therapist-guided internet delivered prolonged exposure with therapist-guided internet delivered cognitive-behavioral therapy The primary outcome is the blind-rater administered Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).

Secondary outcomes are cost effectiveness, mediators of change, dropout rate, and negative effects.

The trial will also be preregistered at the Open Science Framework.

Research questions to be answered are:

1. Is guided i-CBT with exposure more efficacious than an active control condition (therapist-supported internet-delivered psychoeducation, relaxation and support) in regard to reduction of blinded assessor rated PTSD symptom severity 1-month post-treatment?
2. Is guided i-CBT with exposure more cost-effective than an active control condition (therapist-supported internet-delivered psychoeducation, relaxation and support) in regard to reduction of blinded assessor rated PTSD symptom severity 1-month post-treatment?
3. Are the therapeutic gains of i-CBT maintained at long term follow up (6 and 12 months after treatment)?
4. Is guided i-CBT with exposure more efficacious than an active control condition (therapist-supported internet-delivered psychoeducation, relaxation and support) in regard to reduction in depressive symptoms and increase in quality of life up to 12 months after treatment completion?
5. What are the mediators of change in guided i-CBT for PTSD?

ELIGIBILITY:
Inclusion Criteria:

* current primary diagnosis PTSD according to DSM-5 diagnostic criteria
* be 18 years of age or older
* be able to read and communicate fluently in Swedish
* have had a stable dose of any psychotropic medication for at least 4 weeks prior to study entry
* Daily access to a computer or device with internet connection

Exclusion Criteria:

* PTSD is not the primary concern
* Initiation or adjustment of any psychotropic medication within the last 4 weeks prior to commencement of treatment
* Serious mental health symptoms, such as mania, psychosis, alcohol, or substance use disorders or current suicide risk warranting immediate clinical attention.
* Ongoing trauma-focused CBT or Eye movement desensitization and reprocessing therapy
* Ongoing trauma-related threat (e.g. living with a violent spouse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as assessed by the Clinician Administered PTSD Scale (CAPS-5) | Baseline, 1-month (primary endpoint), 6-month and 12-month post-treatment
  The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.

SECONDARY OUTCOMES:
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | Baseline, through the treatment period up to 10 weeks and 1-month, 6-month and 12-month post-treatment]
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in ICD-11 PTSD and complex PTSD symptoms as assessed by the International Trauma Questionnaire (ITQ). | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  The ITQ includes six items measuring each PTSD symptom cluster and these items measure how bothersome each symptom has been in the past month. The ITQ also includes six items measuring each 'Disturbance in Self-Organization' (DSO) symptom in complex PTSD. These items measure how a respondent typically feels, thinks about oneself, and relates to others. The PTSD and DSO symptoms are accompanied by three items measuring associated functional impairments in the domains of social, occupation, and other important areas of life. All items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Thus, PTSD and DSO symptom scores range from 0 to 24 and CPTSD symptom scores range from 0 to 48. Higher scores represents more PTSD and complex PTSD symptoms.
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Change in quality of life measured by Euroqol, EQ-5D | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Change in overall health from baseline to post treatment and follow up . EQ-5D is a standardized self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.
Change in Assessing Quality of Life 6 Dimensions (AQoL-6D) | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Used to assess cost-effectiveness. 20 questions that assess different aspects of quality of life. The AQoL provides a utility score that ranges from 1.00 (full health) to 0.00 (death-equivalent health states) to -0.04 (health states worse than death.
Change in Treatment Inventory of Costs in Psychiatric Patients (TIC-P) | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Self-rated questionnaire on healthcare utilization and productivity losses in patients with a psychiatric disorder. The TIC-P questionnaire measures costs in two dimensions: use of health resources and loss of productivity. Lower cost is better.
Adverse events related to treatment measured by the Negative effects questionnaire | Immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Self-rated questionnaire on negative effects. It contains 32 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances. The total score of the NEQ ranges from 0 to 80 points, a higher score reflects more negative effects.
Participants satisfaction with treatment, assessed by The Client Satisfaction Questionnaire (CSQ-8). | Immediately after treatment completion
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Number of completed treatment modules | Baseline up to treatment completion at 10 weeks
  Data will be gathered on total number of completed modules during the 10 week treatment.
Number of messages sent and received in the digital platform | Baseline up to treatment completion at 10 weeks
  Data will be gathered on total number of messages sent and received back and forth between the participant and the therapist during the 10 week treatment.

OTHER OUTCOMES:
Differences in treatment credibility between arms | After completion of the first treatment module (week 1 from baseline)
  Measures treatment expectancy and rationale credibility. The CEQ is a 5-item measure of the treatment's credibility and the patients' expectations. The patients assess each domain on a 11-point likert scale (scored 0-10), with a total score ranging between 0-50 where higher score indicates higher credibility and higher expectations.
Differences in experience of working alliance between arms | After completion of the third module (week 3 from baseline)
  Measures the therapeutic alliance in therapy. The WAI-SR is a 12-item measure of the patient's experience of their working alliance with the therapist. The patients assess each item on a 7-point likert scale (scored 0-6), with a total score ranging between 0-72 where higher score indicates higher better working alliance according to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bragesjö, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Traumaprogrammet, Psykiatri Sydväst, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bragesjo M, Ivanov VZ, Andersson E, Ruck C. Study protocol of a randomized controlled superiority trial of Huddinge Online Prolonged Exposure therapy (HOPE) for adults with posttraumatic stress disorder. Trials. 2025 Dec 12. doi: 10.1186/s13063-025-09361-0. Online ahead of print. PMID 41388429